CLINICAL TRIAL: NCT02519491
Title: Utility of a Smart Phone Application in Assessing Radial Artery Patency - the CAPITAL iRADIAL Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 20150116-01H
Record Dates: First submitted 2015-08-04; First posted 2015-08-11 (Estimated); Results first posted 2021-05-04 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-10

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Modified Allen's Test (Active Comparator): The Modified Allen's Test to assess radial and ulnar patency.
  Interventions: Other: Modified Allen Test
- Iphone assessment (Active Comparator): iPhone assessment of radial and ulnar patency.
  Interventions: Other: Iphone artery assessment

INTERVENTIONS:
Other: Modified Allen Test — The Modified Allen's Test (MAT) will be performed in a well-lit room on both of the participant's hands. This technique will involve compression of both the radial and ulnar arteries by the investigator to assess patency of the contralateral artery. The participant will then be asked to clench and open their hand several times. The participant will then be asked to maintain their hand in an open position. The investigator will then release the compression over the ulnar artery and observe for palmar blush. The length of time to achieve maximal palmar blush will be recorded. This technique will then be repeated by maintaining compression over the ulnar artery and releasing of the compression over the radial artery.
  Arms: Modified Allen's Test
Other: Iphone artery assessment — The iRADIAL iPhone app (Heart Rate, Azumio software) will be used to assess radial and ulnar artery patency. Briefly, the iPhone camera will be placed over the participant's thumb and patency assessed before and immediately following isolated contralateral artery compression for a maximum of two minutes.
  Arms: Iphone assessment

SUMMARY:
Accessing the arteries of the heart through the blood vessels of the wrist is becoming increasingly popular. By obtaining access via the artery in the arm as opposed to the groin, there is less risk of complications and improved patient satisfaction. However, using the wrist can cause blockage of the artery after the procedure. If there is too little blood flow from a second artery that supplies the hand, this could result in significant injury. Therefore, it is important to test these blood vessels in the wrist prior to having this procedure. The best way to evaluate these arteries involves the use of ultrasounds but this takes a long time and is expensive. Therefore, the artery is usually evaluated with a clinical test known as the modified Allen's test, which relies on the doctor watching the flushing of the hand during compression of the artery. Currently smart phones with cameras are able to assess blood flow by passing light through the skin and watching differences in brightness. This may be a better way to assess the arteries in the hand as it is less subjective than simply watching the flushing of the hand. This study aims to assess the ability of an iPhone application in determining whether there is sufficient blood flow through the arteries of the wrist and comparing it to the clinical test commonly used.

DETAILED DESCRIPTION:
Over the past decade, the transradial approach to cardiac catheterization has emerged as the preferred method of angiography and intervention. There have been several observational and randomized controlled trials which have shown an association between transradial access and reduced risk of bleeding and other vascular complications, increased cost-effectiveness, improved patient satisfaction, and a mortality benefit in high-risk patient populations. However, this technique does carry risks of complications including radial artery occlusion, non-occlusive radial artery injury, radial artery spasm, hand ischemia, pseudoaneurysm, radial artery perforation, nerve damage, arteriovenous fistulisation, and bleeding. Radial artery occlusion is the most commonly noted complication and the clinical impact is unclear. In individuals with intact collateral palmar circulation from the ulnar artery, the individual is usually asymptomatic and do not require further intervention. However, if an individual lacks adequate collateral circulation, that individual is at risk of hand ischemia and loss of tissue or function necessitating surgical intervention or, ultimately, amputation. Thus, it is common practice to assess competency of the collateral palmar circulation prior to transradial cardiac catheterization to mitigate the risks associated with this approach.

The gold standard for assessment of radial artery patency is colour Doppler ultrasound imaging of the artery. This gold standard allows for direct, objective assessment of arterial patency and competency through direct visualization of blood flow. The use of pre-procedural ultrasound remains both labour and resource intensive and hence is not feasible for practical use, therefore a physician must rely on clinical assessment of collateral circulation. This has been traditionally evaluated through use of the modified Allen's test (MAT), a technique performed at the bedside as part of the pre-procedural physical examination. More recently, the introduction of plethysmography and pulse oximetry have been utilized to theoretically provide a more objective measure of assessing collateral circulation, though these too are limited by the available resources. Given the ever increasing prevalence of smart phones, this study aims to address the utility and feasibility of an iPhone application in determining adequacy of collateral palmar circulation. Should this iPhone application provide superior diagnostic accuracy, it could quickly become an alternative method of providing an objective measure of collateral palmar circulation rather than relying on the subjective MAT.

ELIGIBILITY:
Inclusion Criteria:

* All persons who are patients at the University of Ottawa Heart Institute and are candidates for coronary angiography.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2015-07; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Hibbert, MD, PhD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Di Santo P, Harnett DT, Simard T, Ramirez FD, Pourdjabbar A, Yousef A, Moreland R, Bernick J, Wells G, Dick A, Le May M, Labinaz M, So D, Motazedian P, Jung RG, Chandrasekhar J, Mehran R, Chong AY, Hibbert B. Photoplethysmography using a smartphone application for assessment of ulnar artery patency: a randomized clinical trial. CMAJ. 2018 Apr 3;190(13):E380-E388. doi: 10.1503/cmaj.170432. PMID 29615421

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Modified Allen's Test | Iphone Assessment
Started | 219 | 219
Completed | 219 | 219
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population is the same as the assignment in Participant Flow
Groups:
- Total: Total of all reporting groups
Arm/Group | Modified Allen's Test | Iphone Assessment | Total
Number analyzed (Participants) | 219 | 219 | 438
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (13.2) | 67.0 (12.5) | 66.3 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 70 | 153
  Male | 136 | 149 | 285
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 11 | 31
  Not Hispanic or Latino | 199 | 208 | 407
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Accuracy
Description: Diagnostic accuracy of the iRADIAL iPhone application in assessing competency of the collateral blood supply to the hand by comparing the results of the iPhone application to the gold standard (i.e. Doppler ultrasound)
Time Frame: 1 year
Population: Intention to treat
Measure: Number (95% Confidence Interval); unit: Overall diagnostic accuracy (%)
Arm/Group | Modified Allen's Test | Iphone Assessment
Number analyzed (Participants) | 219 | 219
Overall diagnostic accuracy (%) | 81.7 [76.0 to 86.6] | 91.8 [87.3 to 95.1]

ADVERSE EVENTS:
Time Frame: From randomization until discharge from the hospital, up to 1 week
Description: There are no differences in definitions.
Arm/Group | Modified Allen's Test | Iphone Assessment
All-Cause Mortality (participants affected / at risk) | 0/219 | 0/219
Serious Adverse Events (participants affected / at risk) | 0/219 | 0/219
Other Adverse Events (participants affected / at risk) | 0/219 | 0/219

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT02519491/Prot_SAP_000.pdf